CLINICAL TRIAL: NCT00304798
Title: Pilot Study of Admission Versus Discharge After Transient Ischemic Attack (TIA)
Brief Title: Study of Admission Versus Discharge After Transient Ischemic Attack (TIA)
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UCSD IRB #051272
Record Dates: First submitted 2006-03-16; First posted 2006-03-20 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2007-03

CONDITIONS: Transient Ischemic Attack (TIA); Stroke
Keywords: Transient Ischemic Attack (TIA).; Stroke.; Hospital admission.
MeSH Terms: conditions — Ischemic Attack, Transient; Stroke

ARMS (2):
- Admission (Experimental): Admission
  Interventions: Behavioral: Hospital admission
- Discharge (No Intervention): Discharge

INTERVENTIONS:
Behavioral: Hospital admission
  Arms: Admission

SUMMARY:
Evaluate for difference in outcome between hospital admission versus discharge after recent TIA, and evaluate feasibility of a larger study.

DETAILED DESCRIPTION:
20 patients will be randomized within 24 hours of a TIA to be admitted to the hospital or discharged to home, and the investigator will compare outcomes, cost, and evaluate the feasibility of a larger study.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 and older.
* Clinical diagnosis of TIA within 24 hours of consent.

Exclusion Criteria:

* Crescendo TIAs, defined as multiple within 24 hours of presentation.
* Posterior circulation TIAs diagnosed clinically by a member of the Stroke Team.
* High grade carotid stenosis.
* Any compelling medical reason they should or should not be admitted or discharged (for example decompensated congestive heart failure, unstable angina, new EKG changes, pneumonia, sepsis). Patients will only be enrolled if the only consideration for admission is the TIA, and they otherwise meet appropriate standard of care criteria for discharge to home.
* Patients will be excluded if no one can be with them for the next 12 hours to ensure a rapid call to 911 should problems arise, specifically stroke.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-03; Study Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
modified Rankin Scale at one year. | 1 year

SECONDARY OUTCOMES:
Stroke and TIA incidence at one year | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Matt B Jensen, MD, Principal Investigator — UCSD Stroke Center
Locations (1):
- UCSD, San Diego, California, United States